CLINICAL TRIAL: NCT04373863
Title: Let's Get to Know Your Health Better? Assessment of Lifestyle, Blood Pressure and Cholesterol in the Population of Employees Libbs Farmacêutica LTDA.
Brief Title: Assessment of Lifestyle, Blood Pressure, Cholesterol and Glycated Hemoglobin in a Specific Population
Acronym: LB1901
Status: Completed | Type: Observational
Sponsor: Libbs Farmacêutica LTDA (Industry)
Responsible Party: Sponsor
Other Study IDs: LB1901
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2022-07

CONDITIONS: Cholesterol; Lipidosis; Arterial Hypertension; Blood Glucose, High
Keywords: glycated hemoglobin; Cholesterol; Arterial Hypertension; smoking
MeSH Terms: conditions — Lipidoses; Hypertension; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project Shall we get to know your health better? Lifestyle assessment, blood pressure and cholesterol in the population of Libbs Farmacêutica employeesLTDA.; consists of a study that will bring knowledge and enable quantificationof risk factors related to cardiovascular diseases in this population above mentioned.

DETAILED DESCRIPTION:
The social relevance of this study is related to the knowledge and quantification of eating habits and lifestyles related to cardiovascular diseases in the population of employees, also referred to in this document as "employees", from Libbs Farmacêutica Ltda. Based on an observation and statistical analysis of the data obtained in this study, internal policies will be promoted that aim to improve eating habits, physical activity and decrease smoking.

ELIGIBILITY:
Inclusion Criteria:

* Being an employee Libbs Farmacêutica Ltda;

Exclusion Criteria:

* not applicable

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This research project will be conducted during various internal and external institutional events, and in specific actions carried out at Libbs units located in Barra Funda (administrative unit) and in the city of Embu das Artes (production unit).
Sampling Method: Probability Sample
Enrollment: 2472 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Descriptive questionnaire | until December 2020
  Descriptive information about lifestyle and family history and through exams, blood pressure and serum cholesterol values in the population of Libbs Farmacêutica Ltda employees.

SECONDARY OUTCOMES:
Prevalence of hypercholesterolemia and arterial hypertension | until December 2020
  Quantify the prevalence of hypercholesterolemia (serum total cholesterol above 200mg / dL - worst case) and hypertension (systolic blood pressure above 140mmHg or diastolic blood pressure above 90mmHg - worst case)
Glycated hemoglobin (HbA1c) values | until December 2020
  Track the glycated hemoglobin (HbA1c) values of the research participants, in order to know the average blood glucose levels in the last 3 months before the day of the exam and quantify the prevalence of participants who have HbA1c above the value considered normal in literature, which is up to 5.6% (best scenario)
Data correlation | until December 2020
  * Correlate eating habits with socioeconomic characteristics;
  * Correlate the values of serum cholesterol, blood pressure and glycated hemoglobin with eating habits, level of physical activity practiced and prevalence of smoking

CONTACTS AND LOCATIONS:
Locations (1):
- Augusto Theodoro de Figueiredo, São Paulo, Brazil